CLINICAL TRIAL: NCT05063149
Title: Protecting Late-moderate Preterm Infants From Respiratory Tract Infections and Wheeze in Their First Years of Life by Using Bacterial Lysates.
Brief Title: Protecting Preterm Infants From Respiratory Tract Infections and Wheeze by Using Bacterial Lysates.
Acronym: PROTEA
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Franciscus Gasthuis (Other)
Collaborators: Leiden University Medical Center (Other); Maastricht University Medical Center (Other)
Responsible Party: Principal Investigator, Gerdien Tramper, Pediatrician/clinical researcher, principal investigator, Franciscus Gasthuis
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: NL76165.100.20
Record Dates: First submitted 2021-08-24; First posted 2021-09-30 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Wheezing; LRTI; Premature
MeSH Terms: conditions — Respiratory Sounds; Premature Birth | interventions — Broncho-Vaxom

STUDY DESIGN:
Intervention Model Description: Half of the participants (250) will receive treatment (Broncho-Vaxom) and the other half will receive placebo. Randomization will be stratified for gestational age (moderate (30+0-32+6) vs. late (33+0-35+6) prematurity). In the follow-up study Protea-2, infants from the treatment arm in year 1 will be randomised to receive Broncho-Vaxom or placebo in year 2. Randomisation will stratified for gestational age again, but also for the amount of lower respiratory episodes in year 1 (<2 vs. >/=2) Infants from the control arm in year 1 will not receive treatment in year 2.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Study subjects, all study investigators including the principal investigator and treating physicians will be blinded for the allocation during the complete study period. A sealed envelope with the treatment allocation per code is present at the pharmacy to be used only when 1) crucial for a medical emergency, 2) the participant will continue with Protea-2 and the database concerning year 1 is locked for this specific participant, and 3) at trial completion after the last patient last visit.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Broncho-Vaxom treatment (Active Comparator): Infants in this arm will be given 3,5mg bacterial lysate (OM-85) 10 days per month from 6 weeks after birth until 12 months of age.
  At age 12 months they will be (if informed consent for Protea-2 is provided) randomised over Broncho-Vaxom treatment and placebo again.
  Interventions: Drug: Broncho-Vaxom
- Placebo (Placebo Comparator): Infants in this arm will be given a placebo powder from a capsule that will be indistinguishable from the active study drug.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Broncho-Vaxom — Broncho-Vaxom is a bacterial extract comprising lyophilised fractions of 21 different inactivated bacterial strains, which are frequently causing RTI.
  Other Names: OM-85; Broncho-Vaxom concentrate (Bacterial lysate)
  Arms: Broncho-Vaxom treatment
Other: Placebo — Placebo powder from a capsule will be given, which will be indistinguishable from the active study drug.
  Arms: Placebo

SUMMARY:
The primary objective of this study is to reduce respiratory tract infections and wheezing in moderate-late preterms in the first years of life by bacterial lysate administration. Next to determine the correlation of biological markers with respiratory symptoms, immune protection and treatment effect.

DETAILED DESCRIPTION:
This is a randomised placebo-controlled trial including 500 otherwise healthy moderate-late preterm infants. Participants will receive bacterial lysate (OM-85/Broncho-Vaxom, 3,5mg) or placebo powder for ten days each month, from 6-10 weeks after birth until 12 months after birth. At 12 months, parents of participants are asked to join in Protea-2. If they do, participants in the treatment arm of year 1 are randomised again over placebo and OM-85 and treated until the age of 24 months. Clinical data will be continuously collected by e-Health and 3 (possibly digital) study visits; with optional biological sampling and lung function at baseline, 6 and 12 months. And in case of participation in Protea-2 also at 24 months.

Main study parameters are doctor diagnosed lower RTI and wheezing episodes in the first year of life. Biological sampling will allow investigation of immune maturation, as well as microbiome development in the respiratory tract and gut. Also, biomarkers for risk-group selection and/or treatment success will be examined.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age at delivery between 30+0 and 35+6 weeks
* Postnatal age at least 6 weeks at randomization & postmenstrual age at least 37 weeks
* Written informed consent by both parents or formal caregivers

Exclusion Criteria:

* Underlying other severe respiratory disease such as broncho-pulmonary dysplasia (unexpected in this group); hemodynamic significant cardiac disease; immunodefi-ciency; severe failure to thrive; birth asphyxia with predicted poor neurological out-come; syndrome or serious congenital disorder.
* Lower RTI before randomization
* Dysmaturity and/or weight < 2.5 kg at age of randomization.
* Maternal TNF-alpha inhibitors or other immunosuppression during pregnancy and/or breastfeeding
* Parents unable to speak and read Dutch/English language
* Known allergic hypersensitivity to the active ingredients/substance or to any of the excipients.

Ages: 6 Weeks to 10 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 500 (Estimated)
Dates: Start 2022-01-18 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Total number of physician diagnosed lower RTI and wheezing episodes in the first year of life | In the first year of life.
  Recorded by frequent questionnaires

SECONDARY OUTCOMES:
Time to first lower RTI or wheezing episode | In the first and second year of life.
  Recorded by short weekly questionnaires (which will be filled in during the first year of life) and more extensive questionnaires every six months in the first and second year of life.
Total number of RTI | In the first and second year of life.
  Recorded by short weekly questionnaires (which will be filled in during the first year of life) and more extensive questionnaires every six months in the first and second year of life.
Total number of wheezing episodes | In the first and second year of life.
  Recorded by short weekly questionnaires (which will be filled in during the first year of life) and more extensive questionnaires every six months in the first and second year of life.
Distribution of viruses | In the first year of life.
  Viruses present in the nasofarynx during complaints of lower respiratory tract infection or wheezing. Nasofaryngeal swabs will be taken in case of complaints during the first year of life. In the second year of life this will not be done.
Medication use (bronchodilators, corticosteroids, antibiotics) | In the first and second year of life.
  Recorded by short weekly questionnaires (which will be filled in during the first year of life) and more extensive questionnaires every six months in the first and second year of life.
Lung function as measured by expiratory variability index (Ventica) | In the first year of life.
  Measured at age 6-10 weeks (baseline), 6 months and 12 months in a subset of participants.
Quality of life questionnaires | In the first and second year of life.
  Recorded by extensive questionnaires every six months in the first and second year of life.
(serious) adverse events | In the first year of life.
  Will be reported by parents immediately. Respiratory episodes are not regarded as an (S)AE since these episodes comprise primary and secondary outcomes. (S)AE's are only expected in the first year of life because the treatment stops at the age of 12 months.
Serum specific IgE (allergen sensitization) at 12 months | At age 12 months
  Total IgE and house dust mite specific IgE
Infant vaccination titers at 12 months | At age 12 months
  Vaccination titers of haemohilus influenza type B, pneumococci, tetanus
Costs- and cost-effectiveness | In the first and second year of life.
  Estimated from information from standardized questionnaires

OTHER OUTCOMES:
Gut and respiratory microbiome composition | In the first year of life.
  Measured from faeces and nasofaryngeal swabs taken at age 6-10 weeks, 6 months and 12 months.
Secretory IgA in saliva | In the first year of life
  Saliva will be collected at age 6-10 weeks, 6 months and 12 months.
Immune maturation: immune cells in nasal epithelium | In the first year of life
  Collected by nasal scraping at age 6-10 weeks, 6 months and 12 months. Analysed using masscytometry.
Immune maturation: chemokines and cytokines in nasal lining fluid | In the first year of life
  Collected by nasosorption at age 6-10 weeks, 6 months and 12 months. Analysed using Luminex cyto/chemokine assay.
Immune maturation: immune cells in bloodsamples | In the first year of life
  Collected by blooddraws at age 6-10 weeks, 6 months and 12 months. Analysed using masscytometry.
Serum IgE (total and specific to house dust mite) | At age 12 months
  Measured in blood samples which will be drawn at age 12 months
Immune maturation: Single cell transcriptomics | At age 12 months
  Performed on blood drawn at age 12 months
Whole blood stimulation essays | At age 12 months
  Performed on blood drawn at age 12 months
Biomarkers predictive of high morbidity and/or treatment success | In the first year of life.
  From combined microbial and immunological data

CONTACTS AND LOCATIONS:
Locations (1):
- Franciscus Gasthuis & Vlietland, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Researchdata will be shared in data repositories according to the FAIR principle. Clinical data about respiratory health will be shared in the DANS repository. Inlcuding metadata which will ensure reusability. Sequencing data will be shared online in the ENA repository which will provide an unique global identifier. All used bioinformatics pipelines for data analysis will be made accessible on a GitHub account. Immunological data will be shared in NCBI Gene Expression omnibus and ImmPort. Used analysis pipelines for the transcriptomics data will also be tracked and can be shared using a Github account.
  All data shared will be pneudonymized.
Time Frame: Data will come available after publication of the data in articles by initating researchers.
Access Criteria: Data will be available under restricted access. A request for data sharing will include at least the reason for request (for what will the receiver use the data?) and agreements about authorship.

REFERENCES:
- [Background] Haataja P, Korhonen P, Ojala R, Hirvonen M, Korppi M, Gissler M, Luukkaala T, Tammela O. Hospital admissions for lower respiratory tract infections in children born moderately/late preterm. Pediatr Pulmonol. 2018 Feb;53(2):209-217. doi: 10.1002/ppul.23908. Epub 2017 Nov 29. PMID 29193814
- [Background] Pramana IA, Latzin P, Schlapbach LJ, Hafen G, Kuehni CE, Nelle M, Riedel T, Frey U. Respiratory symptoms in preterm infants: burden of disease in the first year of life. Eur J Med Res. 2011 May 12;16(5):223-30. doi: 10.1186/2047-783x-16-5-223. PMID 21719396
- [Background] Vrijlandt EJ, Kerstjens JM, Duiverman EJ, Bos AF, Reijneveld SA. Moderately preterm children have more respiratory problems during their first 5 years of life than children born full term. Am J Respir Crit Care Med. 2013 Jun 1;187(11):1234-40. doi: 10.1164/rccm.201211-2070OC. PMID 23525931
- [Background] Perez-Yarza EG, Moreno-Galdo A, Ramilo O, Rubi T, Escribano A, Torres A, Sardon O, Oliva C, Perez G, Cortell I, Rovira-Amigo S, Pastor-Vivero MD, Perez-Frias J, Velasco V, Torres-Borrego J, Figuerola J, Barrio MI, Garcia-Hernandez G, Mejias A; SAREPREM 3235 investigators. Risk factors for bronchiolitis, recurrent wheezing, and related hospitalization in preterm infants during the first year of life. Pediatr Allergy Immunol. 2015 Dec;26(8):797-804. doi: 10.1111/pai.12414. Epub 2015 Jul 1. PMID 26031206
- [Background] Edwards MO, Kotecha SJ, Lowe J, Richards L, Watkins WJ, Kotecha S. Management of Prematurity-Associated Wheeze and Its Association with Atopy. PLoS One. 2016 May 20;11(5):e0155695. doi: 10.1371/journal.pone.0155695. eCollection 2016. PMID 27203564
- [Background] Kotecha S, Clemm H, Halvorsen T, Kotecha SJ. Bronchial hyper-responsiveness in preterm-born subjects: A systematic review and meta-analysis. Pediatr Allergy Immunol. 2018 Nov;29(7):715-725. doi: 10.1111/pai.12957. Epub 2018 Sep 5. PMID 30014518
- [Background] Moschino L, Carraro S, Baraldi E. Early-life origin and prevention of chronic obstructive pulmonary diseases. Pediatr Allergy Immunol. 2020 Feb;31 Suppl 24:16-18. doi: 10.1111/pai.13157. PMID 32017219
- [Background] Tirone C, Pezza L, Paladini A, Tana M, Aurilia C, Lio A, D'Ippolito S, Tersigni C, Posteraro B, Sanguinetti M, Di Simone N, Vento G. Gut and Lung Microbiota in Preterm Infants: Immunological Modulation and Implication in Neonatal Outcomes. Front Immunol. 2019 Dec 12;10:2910. doi: 10.3389/fimmu.2019.02910. eCollection 2019. PMID 31921169
- [Background] Stewart CJ, Embleton ND, Marrs EC, Smith DP, Nelson A, Abdulkadir B, Skeath T, Petrosino JF, Perry JD, Berrington JE, Cummings SP. Temporal bacterial and metabolic development of the preterm gut reveals specific signatures in health and disease. Microbiome. 2016 Dec 29;4(1):67. doi: 10.1186/s40168-016-0216-8. PMID 28034304
- [Background] Arboleya S, Binetti A, Salazar N, Fernandez N, Solis G, Hernandez-Barranco A, Margolles A, de Los Reyes-Gavilan CG, Gueimonde M. Establishment and development of intestinal microbiota in preterm neonates. FEMS Microbiol Ecol. 2012 Mar;79(3):763-72. doi: 10.1111/j.1574-6941.2011.01261.x. Epub 2011 Dec 15. PMID 22126419
- [Background] Hill CJ, Lynch DB, Murphy K, Ulaszewska M, Jeffery IB, O'Shea CA, Watkins C, Dempsey E, Mattivi F, Tuohy K, Ross RP, Ryan CA, O' Toole PW, Stanton C. Evolution of gut microbiota composition from birth to 24 weeks in the INFANTMET Cohort. Microbiome. 2017 Jan 17;5(1):4. doi: 10.1186/s40168-016-0213-y. PMID 28095889
- [Background] Pattaroni C, Watzenboeck ML, Schneidegger S, Kieser S, Wong NC, Bernasconi E, Pernot J, Mercier L, Knapp S, Nicod LP, Marsland CP, Roth-Kleiner M, Marsland BJ. Early-Life Formation of the Microbial and Immunological Environment of the Human Airways. Cell Host Microbe. 2018 Dec 12;24(6):857-865.e4. doi: 10.1016/j.chom.2018.10.019. Epub 2018 Nov 29. PMID 30503510
- [Background] Carraro S, Scheltema N, Bont L, Baraldi E. Early-life origins of chronic respiratory diseases: understanding and promoting healthy ageing. Eur Respir J. 2014 Dec;44(6):1682-96. doi: 10.1183/09031936.00084114. Epub 2014 Oct 16. PMID 25323240
- [Background] Martinez FD. Childhood Asthma Inception and Progression: Role of Microbial Exposures, Susceptibility to Viruses and Early Allergic Sensitization. Immunol Allergy Clin North Am. 2019 May;39(2):141-150. doi: 10.1016/j.iac.2018.12.001. PMID 30954166
- [Background] Abreo A, Wu P, Donovan BM, Ding T, Gebretsadik T, Huang X, Stone CA, Turi KN, Hartert TV. Infant Respiratory Syncytial Virus Bronchiolitis and Subsequent Risk of Pneumonia, Otitis Media, and Antibiotic Utilization. Clin Infect Dis. 2020 Jun 24;71(1):211-214. doi: 10.1093/cid/ciz1033. PMID 31630167
- [Background] Melville JM, Moss TJ. The immune consequences of preterm birth. Front Neurosci. 2013 May 21;7:79. doi: 10.3389/fnins.2013.00079. eCollection 2013. PMID 23734091
- [Background] McGreal EP, Hearne K, Spiller OB. Off to a slow start: under-development of the complement system in term newborns is more substantial following premature birth. Immunobiology. 2012 Feb;217(2):176-86. doi: 10.1016/j.imbio.2011.07.027. Epub 2011 Jul 30. PMID 21868122
- [Background] Olin A, Henckel E, Chen Y, Lakshmikanth T, Pou C, Mikes J, Gustafsson A, Bernhardsson AK, Zhang C, Bohlin K, Brodin P. Stereotypic Immune System Development in Newborn Children. Cell. 2018 Aug 23;174(5):1277-1292.e14. doi: 10.1016/j.cell.2018.06.045. PMID 30142345
- [Background] Round JL, Mazmanian SK. Inducible Foxp3+ regulatory T-cell development by a commensal bacterium of the intestinal microbiota. Proc Natl Acad Sci U S A. 2010 Jul 6;107(27):12204-9. doi: 10.1073/pnas.0909122107. Epub 2010 Jun 21. PMID 20566854
- [Background] Sjogren YM, Tomicic S, Lundberg A, Bottcher MF, Bjorksten B, Sverremark-Ekstrom E, Jenmalm MC. Influence of early gut microbiota on the maturation of childhood mucosal and systemic immune responses. Clin Exp Allergy. 2009 Dec;39(12):1842-51. doi: 10.1111/j.1365-2222.2009.03326.x. Epub 2009 Sep 3. PMID 19735274
- [Background] Dzidic M, Abrahamsson TR, Artacho A, Bjorksten B, Collado MC, Mira A, Jenmalm MC. Aberrant IgA responses to the gut microbiota during infancy precede asthma and allergy development. J Allergy Clin Immunol. 2017 Mar;139(3):1017-1025.e14. doi: 10.1016/j.jaci.2016.06.047. Epub 2016 Aug 13. PMID 27531072
- [Background] Matias V, San Feliciano L, Fernandez JE, Lapena S, Garrido E, Ardura J, Soga MJ, Aragon MP, Remesal A, Benito F, Andres J, Centeno F, Marugan V, Bachiller R, Bermejo-Martin JF. Host and environmental factors influencing respiratory secretion of pro-wheezing biomarkers in preterm children. Pediatr Allergy Immunol. 2012 Aug;23(5):441-7. doi: 10.1111/j.1399-3038.2012.01269.x. Epub 2012 May 3. PMID 22554061
- [Background] Teo SM, Mok D, Pham K, Kusel M, Serralha M, Troy N, Holt BJ, Hales BJ, Walker ML, Hollams E, Bochkov YA, Grindle K, Johnston SL, Gern JE, Sly PD, Holt PG, Holt KE, Inouye M. The infant nasopharyngeal microbiome impacts severity of lower respiratory infection and risk of asthma development. Cell Host Microbe. 2015 May 13;17(5):704-15. doi: 10.1016/j.chom.2015.03.008. Epub 2015 Apr 9. PMID 25865368
- [Background] Thorsen J, Rasmussen MA, Waage J, Mortensen M, Brejnrod A, Bonnelykke K, Chawes BL, Brix S, Sorensen SJ, Stokholm J, Bisgaard H. Infant airway microbiota and topical immune perturbations in the origins of childhood asthma. Nat Commun. 2019 Nov 1;10(1):5001. doi: 10.1038/s41467-019-12989-7. PMID 31676759
- [Background] Vissing NH, Larsen JM, Rasmussen MA, Chawes BL, Thysen AH, Bonnelykke K, Brix S, Bisgaard H. Susceptibility to Lower Respiratory Infections in Childhood is Associated with Perturbation of the Cytokine Response to Pathogenic Airway Bacteria. Pediatr Infect Dis J. 2016 May;35(5):561-6. doi: 10.1097/INF.0000000000001092. PMID 26910587
- [Background] Blanken MO, Rovers MM, Molenaar JM, Winkler-Seinstra PL, Meijer A, Kimpen JL, Bont L; Dutch RSV Neonatal Network. Respiratory syncytial virus and recurrent wheeze in healthy preterm infants. N Engl J Med. 2013 May 9;368(19):1791-9. doi: 10.1056/NEJMoa1211917. PMID 23656644
- [Background] Luoto R, Ruuskanen O, Waris M, Kalliomaki M, Salminen S, Isolauri E. Prebiotic and probiotic supplementation prevents rhinovirus infections in preterm infants: a randomized, placebo-controlled trial. J Allergy Clin Immunol. 2014 Feb;133(2):405-13. doi: 10.1016/j.jaci.2013.08.020. Epub 2013 Oct 13. PMID 24131826
- [Background] Niele N, van Zwol A, Westerbeek EA, Lafeber HN, van Elburg RM. Effect of non-human neutral and acidic oligosaccharides on allergic and infectious diseases in preterm infants. Eur J Pediatr. 2013 Mar;172(3):317-23. doi: 10.1007/s00431-012-1886-2. Epub 2012 Nov 7. PMID 23132642
- [Background] Pfefferle PI, Prescott SL, Kopp M. Microbial influence on tolerance and opportunities for intervention with prebiotics/probiotics and bacterial lysates. J Allergy Clin Immunol. 2013 Jun;131(6):1453-63; quiz 1464. doi: 10.1016/j.jaci.2013.03.020. Epub 2013 May 2. PMID 23643095
- [Background] Yin J, Xu B, Zeng X, Shen K. Broncho-Vaxom in pediatric recurrent respiratory tract infections: A systematic review and meta-analysis. Int Immunopharmacol. 2018 Jan;54:198-209. doi: 10.1016/j.intimp.2017.10.032. Epub 2017 Nov 16. PMID 29154122
- [Background] Cazzola M, Anapurapu S, Page CP. Polyvalent mechanical bacterial lysate for the prevention of recurrent respiratory infections: a meta-analysis. Pulm Pharmacol Ther. 2012 Feb;25(1):62-8. doi: 10.1016/j.pupt.2011.11.002. Epub 2011 Nov 27. PMID 22155205
- [Background] Razi CH, Harmanci K, Abaci A, Ozdemir O, Hizli S, Renda R, Keskin F. The immunostimulant OM-85 BV prevents wheezing attacks in preschool children. J Allergy Clin Immunol. 2010 Oct;126(4):763-9. doi: 10.1016/j.jaci.2010.07.038. PMID 20920766
- [Background] Esposito S, Bianchini S, Bosis S, Tagliabue C, Coro I, Argentiero A, Principi N. A randomized, placebo-controlled, double-blinded, single-centre, phase IV trial to assess the efficacy and safety of OM-85 in children suffering from recurrent respiratory tract infections. J Transl Med. 2019 Aug 23;17(1):284. doi: 10.1186/s12967-019-2040-y. PMID 31443716
- [Background] de Boer GM, Zolkiewicz J, Strzelec KP, Ruszczynski M, Hendriks RW, Braunstahl GJ, Feleszko W, Tramper-Stranders GA. Bacterial lysate therapy for the prevention of wheezing episodes and asthma exacerbations: a systematic review and meta-analysis. Eur Respir Rev. 2020 Nov 27;29(158):190175. doi: 10.1183/16000617.0175-2019. Print 2020 Dec 31. PMID 33246991
- [Background] Sly PD, Galbraith S, Islam Z, Holt B, Troy N, Holt PG. Primary prevention of severe lower respiratory illnesses in at-risk infants using the immunomodulator OM-85. J Allergy Clin Immunol. 2019 Sep;144(3):870-872.e11. doi: 10.1016/j.jaci.2019.05.032. Epub 2019 Jun 8. No abstract available. PMID 31185221
- [Background] Lau S, Gerhold K, Zimmermann K, Ockeloen CW, Rossberg S, Wagner P, Sulser C, Bunikowski R, Witt I, Wauer J, Beschorner J, Menke G, Hamelmann E, Wahn U. Oral application of bacterial lysate in infancy decreases the risk of atopic dermatitis in children with 1 atopic parent in a randomized, placebo-controlled trial. J Allergy Clin Immunol. 2012 Apr;129(4):1040-7. doi: 10.1016/j.jaci.2012.02.005. PMID 22464674
- [Background] Esposito S, Marchisio P, Prada E, Daleno C, Porretti L, Carsetti R, Bosco A, Ierardi V, Scala A, Principi N. Impact of a mixed bacterial lysate (OM-85 BV) on the immunogenicity, safety and tolerability of inactivated influenza vaccine in children with recurrent respiratory tract infection. Vaccine. 2014 May 7;32(22):2546-52. doi: 10.1016/j.vaccine.2014.03.055. Epub 2014 Mar 26. PMID 24681270
- [Background] Seppa VP, Paassilta M, Kivisto J, Hult A, Viik J, Gracia-Tabuenca J, Karjalainen J. Reduced expiratory variability index (EVI) is associated with controller medication withdrawal and symptoms in wheezy children aged 1-5 years. Pediatr Allergy Immunol. 2020 Jul;31(5):489-495. doi: 10.1111/pai.13234. Epub 2020 Mar 17. PMID 32068911
- [Background] de Ruiter K, Jochems SP, Tahapary DL, Stam KA, Konig M, van Unen V, Laban S, Hollt T, Mbow M, Lelieveldt BPF, Koning F, Sartono E, Smit JWA, Supali T, Yazdanbakhsh M. Helminth infections drive heterogeneity in human type 2 and regulatory cells. Sci Transl Med. 2020 Jan 1;12(524):eaaw3703. doi: 10.1126/scitranslmed.aaw3703. PMID 31894102
- [Background] Jochems SP, de Ruiter K, Solorzano C, Voskamp A, Mitsi E, Nikolaou E, Carniel BF, Pojar S, German EL, Reine J, Soares-Schanoski A, Hill H, Robinson R, Hyder-Wright AD, Weight CM, Durrenberger PF, Heyderman RS, Gordon SB, Smits HH, Urban BC, Rylance J, Collins AM, Wilkie MD, Lazarova L, Leong SC, Yazdanbakhsh M, Ferreira DM. Innate and adaptive nasal mucosal immune responses following experimental human pneumococcal colonization. J Clin Invest. 2019 Jul 30;129(10):4523-4538. doi: 10.1172/JCI128865. PMID 31361601
- [Background] Beyrend G, Stam K, Hollt T, Ossendorp F, Arens R. Cytofast: A workflow for visual and quantitative analysis of flow and mass cytometry data to discover immune signatures and correlations. Comput Struct Biotechnol J. 2018 Oct 24;16:435-442. doi: 10.1016/j.csbj.2018.10.004. eCollection 2018. PMID 30450167
- [Background] Galazzo G, van Best N, Bervoets L, Dapaah IO, Savelkoul PH, Hornef MW; GI-MDH consortium; Lau S, Hamelmann E, Penders J. Development of the Microbiota and Associations With Birth Mode, Diet, and Atopic Disorders in a Longitudinal Analysis of Stool Samples, Collected From Infancy Through Early Childhood. Gastroenterology. 2020 May;158(6):1584-1596. doi: 10.1053/j.gastro.2020.01.024. Epub 2020 Jan 18. PMID 31958431
- [Background] Badurdeen S, Marshall A, Daish H, Hatherill M, Berkley JA. Safety and Immunogenicity of Early Bacillus Calmette-Guerin Vaccination in Infants Who Are Preterm and/or Have Low Birth Weights: A Systematic Review and Meta-analysis. JAMA Pediatr. 2019 Jan 1;173(1):75-85. doi: 10.1001/jamapediatrics.2018.4038. PMID 30476973
- [Background] Stein MM, Hrusch CL, Gozdz J, Igartua C, Pivniouk V, Murray SE, Ledford JG, Marques Dos Santos M, Anderson RL, Metwali N, Neilson JW, Maier RM, Gilbert JA, Holbreich M, Thorne PS, Martinez FD, von Mutius E, Vercelli D, Ober C, Sperling AI. Innate Immunity and Asthma Risk in Amish and Hutterite Farm Children. N Engl J Med. 2016 Aug 4;375(5):411-421. doi: 10.1056/NEJMoa1508749. PMID 27518660
- [Background] Karaca NE, Gulez N, Aksu G, Azarsiz E, Kutukculer N. Does OM-85 BV prophylaxis trigger autoimmunity in IgA deficient children? Int Immunopharmacol. 2011 Nov;11(11):1747-51. doi: 10.1016/j.intimp.2011.06.009. Epub 2011 Jul 21. PMID 21771668